CLINICAL TRIAL: NCT05531383
Title: Effect of Early Memantine Administration on Outcome of Patients With Moderate to Severe Traumatic Brain Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Shady Nemr Youssef, Principal investigator, Minia University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 140-2021
Record Dates: First submitted 2022-03-08; First posted 2022-09-08 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Memantine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (group 1) (No Intervention): Patients in the control group (group 1) No memantine administration
- Treatment group (group 2) (Active Comparator): in addition to the standard treatment, they will receive memantine (30 mg) twice daily, either orally or through a nasogastric tube for 7 days, starting on the first day of admission to the hospital. The memantine dose administered in our study was based on the maximum dose of 60 mg/day reported in prior human studies
  Interventions: Drug: Memantine Hydrochloride

INTERVENTIONS:
Drug: Memantine Hydrochloride — study the effect of memantine on platelet, platelet/lymphocyte ratio (PLR) and C reactive protein (CRP) & serum NSE levels in patients with moderate to severe TBI as well as their outcome.
  Other Names: Namenda
  Arms: Treatment group (group 2)

SUMMARY:
Effect of Early Memantine Administration on Outcome of Participents with Moderate to Severe Traumatic Brain Injury

DETAILED DESCRIPTION:
Studying the effect of memantine on platelet, platelet/lymphocyte ratio (PLR) and C reactive protein (CRP) & serum NSE levels in participents with moderate to severe TBI as well as outcome.

Investigators evaluate prognostic effect of memantine on participents with moderate to severe TBI. also to estimate which of platelet, platelet/lymphocyte ratio (PLR), C reactive protein (CRP) or serum NSE levels will be affected by administration of memantine in participents with moderate to severe TBI as a predictor of outcome.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe closed TBI with initial GCS of 4-12
* Age from 18 to 65 years of both sexes
* Able to tolerate enteral feeding and drug administration within the first 24 hours of TBI.

Exclusion Criteria:

* Open TBI or patients who would need open craniotomy later on.
* Comorbid illnesses, such as diabetes mellitus, ischemic heart disease, acute myocardial infarction within the past 48 hours, acute or chronic renal insufficiency, hepatic diseases, autoimmune abnormalities, history of epileptic fits and known malignancies.

Patients with chest, cardiac, abdominal trauma or any other trauma requiring mechanical ventilation.

Patients with body mass index (BMI) <18.5 or > 34.9 kg/m2.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-11-26 (Actual); Primary Completion 2023-11-20 (Estimated); Study Completion 2024-07-09 (Estimated)

PRIMARY OUTCOMES:
prognosis of moderate to sever head injury | 7days
  Evaluating the effect of memantine administration on the conscious level of patients using the Glasgow coma scale

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim Talaat, MD, Study Chair — Minia University
Locations (1):
- Faculty of medecine, Minya, Minya Governorate, Egypt